CLINICAL TRIAL: NCT06492109
Title: The Peripheral Blood Multi-Omics Study on the Association of Sleep Loss With Aging and Alzheimer's Disease
Brief Title: The Peripheral Blood Multi-Omics Study on Sleep Loss
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: First Affiliated Hospital of Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: Multi-omics in Sleep loss
Record Dates: First submitted 2024-06-26; First posted 2024-07-09 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Sleep Deprivation; Aging; Alzheimer Disease; Healthy Lifestyle; Cognitive Decline; Shift-work Disorder
Keywords: sleep loss; multi-omics; Metabolome; aging; alzheimer's disease
MeSH Terms: conditions — Sleep Deprivation; Alzheimer Disease; Cognitive Dysfunction

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Healthy participants (Other): Overall good health, with a BMI between 17 and 26; aged between 18 and 80 years; no complaints of cognitive impairment, normal neurological examination; signed informed consent form.
  Interventions: Behavioral: Sleep manipulation
- Patients with mild cognitive impairment (MCI) (No Intervention): Meets Petersen et al.'s diagnostic criteria for MCI: presence of subjective memory complaints; objective episodic memory impairment (scores on clinical memory tests falling 1-1.5 standard deviations below age- and education-adjusted norms); overall cognitive function is essentially normal, with a score of MMSE ≥ 24 indicating normal cognitive function according to the dementia screening standards specified by the Beijing Collaborative Group; CDR-global score = 0.5; daily living abilities are largely intact (capable of using public transportation, shopping, and managing finances). Does not meet the criteria for dementia according to the International Classification of Diseases, 10th edition (research version), or the National Institute of Neurological and Communicative Disorders and Stroke-Alzheimer's Disease and Related Disorders Association (NINCDS-ADRDA) criteria for probable Alzheimer's disease. Signed informed consent form.
- Patients with Alzheimer's disease (AD) (No Intervention): Meets the NINCDS-ADRDA criteria for probable Alzheimer's disease; CDR-global score = 1; overall cognitive decline: MMSE score of 20-24; impaired daily living abilities: Activities of Daily Living (ADL) scale score > 26. Signed informed consent form.

INTERVENTIONS:
Behavioral: Sleep manipulation — This study will collect the MMSE results as a supplement to the MoCA. The sleep status of subjects will be screened using the Morningness-Eveningness Questionnaire (MEQ), Pittsburgh Sleep Quality Index (PSQI), and Epworth Sleepiness Scale (ESS).
  Subjects must maintain regular sleep and diet before sample collection. Peripheral blood samples will be taken the day before, the day of, and the day after acute sleep deprivation, whether experimentally induced (controlled) or naturally occurring (passive), along with assessment scales including anxiety and depression assessments.
  For chronic sleep deprivation (≥7 days), blood samples will be collected before and after the deprivation period, with anxiety, depression, and cognitive assessments.
  Experimentally induced sleep deprivation takes place under controlled laboratory conditions, whereas passive sleep deprivation arises from external factors such as aging or shift work.
  Arms: Healthy participants

SUMMARY:
Sleep plays a role in cognitive processes such as memory processing, attention processing, and overall cognitive function. In recent years, the bidirectional relationship between sleep loss and aging, as well as related neurodegenerative diseases, has garnered widespread attention. Sleep disorders are a typical clinical manifestation of neurodegenerative diseases such as Alzheimer's disease (AD) and Parkinson's disease and are closely related to the progression of these diseases. However, current research has yet to fully elucidate the physiological responses to sleep loss across different ages and cognitive levels, as well as the association and molecular basis between sleep loss, aging, and neurodegenerative diseases. This study aims to comprehensively characterize the transcriptional and metabolic changes in peripheral blood under sleep loss in populations of different ages and cognitive levels using multi-omics approaches and to preliminarily explore the role of sleep loss in aging and AD.

DETAILED DESCRIPTION:
Participants meeting inclusion and exclusion criteria will include healthy subjects, MCI patients, and AD patients. General information such as age, gender, education level, medical history, family history, medication history, and surgical history will be collected. Cognitive assessments and sleep condition screenings will be conducted, with blood samples collected before and after sleep loss, and anxiety and depression scales administered. Blood samples will be processed using standardized methods for multi-omics analysis. Joint analyses with cognitive levels and sleep conditions will be performed to identify molecular biomarkers associated with age, cognitive levels, and key biological processes related to sleep loss, revealing its association with aging and AD.

This study includes an intervention component, in which part of the participants will undergo controlled (active) or naturally occurred (passive) sleep manipulation (including normal sleep, sleep deprivation, and recovery sleep), as described in the arms and interventions sections. Active sleep deprivation is conducted under controlled experimental conditions, whereas passive deprivation results from natural factors such as age or shift work. Therefore, this study qualifies as a Basic Experimental Study Involving Humans (BESH), as it does not involve the administration of any medicinal product or therapeutic intervention. According to the NIH's four defining questions for BESH:

1. Does the study involve human participants? Yes. This study involves human.
2. Are the participants prospectively assigned to an intervention? Yes. Part of the participants will prospectively assigned to a sequence of controlled sleep conditions (normal sleep, sleep deprivation, and recovery sleep) to investigate related physiological responses.
3. Is the study designed to evaluate the effect of the intervention on the participants? Yes. The aim was to investigate how changes in sleep status affected peripheral blood metabolic and immune phenotypes, as well as behavioral assessments. These served as dependent variables in the analysis.
4. Is the effect being evaluated a health-related biomedical or behavioral outcome? Yes. The outcomes are health related biomedical effects relevant to understanding physiological adaptation, though not intended for clinical application or therapeutic benefit.

In brief, this study involved a part of single arm, non-masked, non-randomized, basic science intervention. These sleep manipulations were transient, reversible, and/or physiologically benign procedures designed to investigate normal biological function.The metabolic and immune phenotype as well as behavioral assessment results were the primary outcome measure of the BESH intervention.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent form；
2. Meet the inclusion criteria for each arms.

Exclusion Criteria:

1. Failure to provide informed consent;
2. Inability to follow study procedures due to issues such as language barriers or cognitive impairment;
3. Regular use of medications that may alter the relationship between sleep and outcome variables (e.g., opioid medications, benzodiazepines, and Z drugs [non-benzodiazepine hypnotics]);
4. History of alcohol abuse, substance abuse, consciousness disorders, cerebrovascular disease, head injury, epilepsy, encephalitis, or other neurological disorders;
5. Diagnosis of schizophrenia, severe depression, anxiety disorders, or other severe psychiatric conditions;
6. Presence of severe arrhythmias, myocardial infarction within the last 6 months, severe pulmonary dysfunction, renal or hepatic insufficiency, severe anemia, severe gastrointestinal diseases, tumors, or other severe medical conditions.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-06-20 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Hamilton Anxiety Rating Scale (HAM-A) | through study completion, an average of 1 month
  The scale consists of 14 items, each defined by a series of symptoms, and measures both psychic anxiety (mental agitation and psychological distress) and somatic anxiety (physical complaints related to anxiety). Each of the 14 items contains a number of symptoms, and each group of symptoms is rated on a scale of zero to four, with four being the most severe. All of these scores are used to compute an overarching score that indicates a person's anxiety severity.
Hamilton Depression Rating Scale (HDRS) | through study completion, an average of 1 month
  The Hamilton Depression Rating Scale (HDRS) is the most commonly used instrument for assessing symptoms of depression. It has been used in many key studies of depression and its treatment. The instrument is designed to be administered by clinicians after a structured or unstructured interview of the patient to determine their symptoms. A total score is calculated by summing the individual scores from each question.
  Scores below 7 generally represent the absence or remission of depression. Scores between 7-17 represent mild depression Scores between 18-24 represent moderate depression Scores 25 and above represent severe depression
Mini-Mental State Examination (MMSE) | through study completion, an average of 1 month
  The Mini Mental State Examination (MMSE) is a tool that can be used to systematically and thoroughly assess mental status. It is an 11-question measure that tests five areas of cognitive function: orientation, registration, attention and calculation, recall, and language. The maximum score is 30. A score of 23 or lower is indicative of cognitive impairment. The MMSE takes only 5-10 minutes to administer and is therefore practical to use repeatedly and routinely.
Montreal Cognitive Assessment (MoCA) | through study completion, an average of 1 month
  The Montreal Cognitive Assessment (MOCA) was initially developed as a test for mild cognitive impairment, but has also been determined to match qualities of the MMSE.80 It assesses seven areas of cognition for a total possible score of 30 points. A score of 25 or less is indicative of cognitive impairment.
Transcriptomic profile | through study completion, an average of 1 month
  A comprehensive transcriptomic from plasma was obtained using RNA sequencing
Metabolic profiling | through study completion, an average of 1 month
  A comprehensive metabolic profile from plasma was obtained using targeted metabolomics analysis and untargeted and targeted lipidomics analysis.
Self reported scales | through study completion, an average of 1 year
  Participants underwent sleep manipulations should report their physical and mental discomforts and score them.

CONTACTS AND LOCATIONS:
Overall Officials: Benyan Luo, Principal Investigator — Zhejiang University
Locations (1):
- The First Affiliated Hospital of Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) is not available to other researchers